CLINICAL TRIAL: NCT03576846
Title: The Effect of Spinal Manipulative Therapy on Heart Rate Variability and Pain, and the Predictive Value of Conditioned Pain Modulation
Brief Title: Spinal Pain and Autonomic Responses to Chiropractic Care
Acronym: SPARC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: University of Southern Denmark (Other)
Responsible Party: Principal Investigator, Iben Axen, Associate Professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KIIMMIIRIA
Record Dates: First submitted 2018-06-20; First posted 2018-07-03 (Actual); Results first posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Neck Pain
Keywords: neck pain; spinal manipulative therapy; heart rate variability; conditioned pain modulation
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized into two arms: 1: stretching exercises only, 2: stretching exercises and Spinal Manipulative Therapy
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The subject will not know the content of the other arm. The care provider cannot be blinded, as he/she will be performing the treatment. The investigator performing the measurements will not be aware of the treatment allocation, and the analyses will be masked for group allocation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Stretching and Spinal Manipulative Therapy
  Interventions: Other: Stretching and Spinal manipulative therapy
- Comparator (Active Comparator): Stretching
  Interventions: Other: Stretching

INTERVENTIONS:
Other: Stretching and Spinal manipulative therapy — Subjects will be instructed to perform a series of progressively difficult stretching exercises for the neck and upper back muscles. In addition, subjects will be treated with Spinal manipulative therapy
  Arms: Intervention
Other: Stretching — Subjects will be instructed to perform a series of progressively difficult stretching exercises for the neck and upper back muscles.
  Arms: Comparator

SUMMARY:
This randomized, single-blinded study will investigate the effects of Spinal Manipulative Therapy on Heart Rate Variability and Pain Sensitivity in a population of patients with recurrent and persistent neck pain. Alongside, the study will also develop a clinical test for Conditioned Pain Modulation and investigate its predictive properties.

DETAILED DESCRIPTION:
Previously, Spinal Manipulative Therapy (SMT) was thought to mechanically affect the restoration of muscular and joint function, by normalising muscle tension and joint mobility. However, recent research has suggested that SMT may be influencing the incoming/ascending pain signals and/or the excitability of the central pain regulating mechanisms. People with chronic neck/shoulder pain have been found to have a disturbance of the Autonomic Nervous System (ANS). Little is known about the changes in the ANS and its relation to changes in pain in a series of treatments conducted in a clinical setting.

This multicentre randomized controlled clinical trial will be carried out in multimodal primary care clinics where both physiotherapists and chiropractors are consulted for musculoskeletal issues are selected to minimize selection bias from the patient's pre-desired treatment modality.

The subjects will be recruited among patients seeking care for persistent or recurrent Neck pain (NP), either self-selected or through referrals from general practitioners in the local areal. The aim is to study the effect of SMT and stretching exercises compared to stretching exercises alone, two well-known interventions for NP, during a two-week treatment regimen.

The primary outcome is the activity of the autonomic nervous system (Heart Rate Variability (HRV), but also Conditioned Pain Modulation (CPM) will be measured. HRV and CPM will be measured at baseline, prior to the third treatment and after the fourth treatment.

The subjective pain experience will be investigated by using two different instruments accessing pain intensity and the affective quality of pain, asked at the assessments during the two weeks of treatment and 2 months after the period of intervention ends.

Highly structured data collection procedures should provide reliable data to answer these questions. The study utilizes normal clinical procedures, which should aid the transferability of the results.

ELIGIBILITY:
Inclusion Criteria:

* minimum 18 years,
* able to read and understand Swedish,
* persistent or recurrent Neck Pain (duration of current episode more than 6 months and at least one previous episode of NP),
* no chiropractic treatment during the previous 3 months.

Exclusion Criteria:

* conditions or medications that will affect the Heart Rate Variability measurements (cardiovascular disease, diabetes, pregnancy, obesity, currently using pain-reducing medication, steroids or antidepressants),
* all contraindications to manual treatment, (anything that could seriously aggravate the pain (such as inflammatory conditions) or signal cerebrovascular injuries (previous drop attacks or a recent episode of new headache or dizziness).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2019-01-04 (Actual); Primary Completion 2020-05-02 (Actual); Study Completion 2020-05-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Iben Axén, Principal Investigator — Karolinska Institutet
Locations (2):
- Sweden (2):
  - Karolinska Institutet, Stockholm
  - Danvik Kiropraktik och Rehab, Stockholm

IPD SHARING:
Plan to Share IPD: No
Anonymized information may be shared with other researchers upon request, pending ethical approval.

REFERENCES:
- [Derived] Galaasen Bakken A, Eklund A, Oksanen A, Axen I. The response to individualized treatment after a standardized treatment protocol among neck pain sufferers: a secondary analysis of a randomized controlled trial. Chiropr Man Therap. 2025 Apr 11;33(1):13. doi: 10.1186/s12998-025-00579-y. PMID 40217263
- [Derived] Bakken AG, Eklund A, Warnqvist A, O'Neill S, Hallman DM, Axen I. Are changes in pain associated with changes in heart rate variability in patients treated for recurrent or persistent neck pain? BMC Musculoskelet Disord. 2022 Oct 4;23(1):895. doi: 10.1186/s12891-022-05842-4. PMID 36192738
- [Derived] Galaasen Bakken A, Eklund A, Hallman DM, Axen I. The effect of spinal manipulative therapy and home stretching exercises on heart rate variability in patients with persistent or recurrent neck pain: a randomized controlled trial. Chiropr Man Therap. 2021 Nov 29;29(1):48. doi: 10.1186/s12998-021-00406-0. PMID 34844625
- [Derived] Bakken AG, Eklund A, Warnqvist A, O'Neill S, Axen I. The effect of two weeks of spinal manipulative therapy and home stretching exercises on pain and disability in patients with persistent or recurrent neck pain; a randomized controlled trial. BMC Musculoskelet Disord. 2021 Oct 27;22(1):903. doi: 10.1186/s12891-021-04772-x. PMID 34706706
- [Derived] Galaasen Bakken A, Axen I, Eklund A, O'Neill S. The effect of spinal manipulative therapy on heart rate variability and pain in patients with chronic neck pain: a randomized controlled trial. Trials. 2019 Oct 12;20(1):590. doi: 10.1186/s13063-019-3678-8. PMID 31606042

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention | Comparator
Started | 66 | 65
Responders | 27 | 26
Non-responders | 27 | 25
Completed | 54 | 41
Not Completed | 12 | 24

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Comparator | Total
Number analyzed (Participants) | 66 | 65 | 131
Age, Continuous [Mean (Standard Deviation); unit: Years] | 57 (14) | 57.5 (36) | 57.2 (13.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 36 | 73
  Male | 29 | 29 | 58
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Heart rate variability [Mean (Standard Deviation); unit: ms] — The reported measure is the RMSSD, Root mean squared successive diferences, recorded with a sampling rate of 1000 Hz between inter-beat-intervals, measured in ms. Population: A few participants did not have HRV measurements of sufficient quality, and their measurements had to be excluded
  ms
    number analyzed (Participants) | 62 | 58 | 120
    (all) | 27 (29) | 29 (21) | 28 (25)

OUTCOME MEASURES:

1. Primary Outcome: Change in Heart Rate Variability
Description: The variation in beat-to-beat heart rate is an indicator of parasympathetic and sympathetic modulation of the heart rhythm. It is measured as the time between two R-waves on the ECG and measured in ms.
Time Frame: 2 weeks, the change is reported between baseline-2 weeks
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | Intervention | Comparator
Number analyzed (Participants) | 62 | 61
ms | 843 (129) | 887 (138)

2. Secondary Outcome: Change in Conditioned Pain Modulation, Measured as the Difference in Pain Intensity Between Two Conditions .
Description: Conditioned Pain Modulation is assessed using a thumb clamp and a cold pressor test. Pain is rated on the Numeric Rating Scale, ranging from 10 (unbearable pain) to 0 (no pain). The outcome is the difference between these two measurements.
Time Frame: The test is done at baseline and again at 2 weeks, and the outcome is the difference between these two scores
Population: In this analysis, the original study arms were not used, and the participants were treated as one cohort.
Measure: Mean (Standard Deviation); unit: NRS change score
Groups:
- Clinical Responders: clinical responders were defined on the basis of changes in clinical neck pain intensity as reported using a reduction of two or more NRS points on a 0-10 scale, between baseline and two-week follow-up (end of the intervention period).
- Clinical non-responders: clinical non-responders were defined on the basis of changes in clinical neck pain intensity as reported between baseline and two-week follow-up (end of the intervention period) where an increase in pain or a reduction of less than two on a numeric rating scale (NRS-11)was considered a clinical non-responder
Arm/Group | Clinical Responders | Clinical non-responders
Number analyzed (Participants) | 53 | 52
NRS change score | -3.3 (0.2) | 0.2 (0.2)

3. Other Pre Specified Outcome: Change in Pain Intensity
Description: Self-reported, using the Numeric Rating Scale (0-10). High scores indicate more severe pain. The outcome is the difference between the scores measured at baseline at at two weeks.
Time Frame: 2 weeks, pain intensity is assessed at Baseline and after 2 weeks, the outcome is the difference between them.
Population: This is an intention-to-treat analysis. Participants are analyzed according to the arm in which they were randomized.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Comparator
Number analyzed (Participants) | 65 | 64
score on a scale | 1.1 (2.085) | 1.1 (2.101)

4. Other Pre Specified Outcome: Change in Disability Score
Description: Neck Disability Index (10 questions, answer options 1-6, summary score, higher score indicating higher disabiity), reported at baseline and at 2 weeks follow up. The measure is the difference between these two scores
Time Frame: 2 weeks
Population: The disability score is based on the instrument Neck Disability Index, and the change is the difference between the last and first measurement, 2 weeks apart
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Comparator
Number analyzed (Participants) | 57 | 58
score on a scale | -2.1 (4.58) | -1.9 (4.21)

5. Other Pre Specified Outcome: Common Side-effects
Description: Description and count of common side effects, data collected through a single question using text messages.
  Thus, the participants described their side-effects, which were categorized and counted.
Time Frame: 1 week
Population: Description and count of side-effects
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Comparator
Number analyzed (Participants) | 66 | 65
Participants | 3 | 1

ADVERSE EVENTS:
Time Frame: The participants were asked to report adverse events 1 day after the first treatment was administered.
Description: Subjects were asked to report any adverse reactions to the first treatment through a text message, i.e. increased tenderness or fatigue in the neck, answered with an NRS-11 scale anchored by the descriptors 'No reaction' (0) and 'Worst reaction imaginable'
Arm/Group | Intervention | Comparator
All-Cause Mortality (participants affected / at risk) | 0/66 | 0/65
Serious Adverse Events (participants affected / at risk) | 0/66 | 0/65
Other Adverse Events (participants affected / at risk) | 3/66 | 1/65
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention (N=66) | Comparator (N=65)
Minor (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1) — Increased pain and discomfort

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The agreement stipulates that the funder has no say in the analysis, interpretation, publication or communication of the results.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-20): https://cdn.clinicaltrials.gov/large-docs/46/NCT03576846/Prot_SAP_000.pdf